CLINICAL TRIAL: NCT01537458
Title: Long-term Outcome After Isolated Tricuspid Valve Repair
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Agency for Science, Technology and Research (Other)
Responsible Party: Sponsor
Other Study IDs: Is_TVR_1
Record Dates: First submitted 2012-02-13; First posted 2012-02-23 (Estimated); Last update posted 2023-01-27 (Actual); Status verified 2012-02

CONDITIONS: Tricuspid Valve Insufficiency
MeSH Terms: conditions — Tricuspid Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Isolated TI repair: Patients that underwent isolated tricuspid valve repair
  Interventions: Procedure: follow-up of isolated tricuspid valve repair

INTERVENTIONS:
Procedure: follow-up of isolated tricuspid valve repair — follow-up of patients that underwent TV repair in the past.

SUMMARY:
Tricuspid valve insufficiency (TI) is often noted on echocardiography. Although severe TI is known to cause significant morbidity and mortality, no good guidelines are available to guide intervention. Literature is mostly confined to tricuspid valve repair concomitant with mitral valve repair. Treatment options for isolated repair have not been investigated thoroughly.

The investigators want to evaluate retrospectively the outcome of isolated tricuspid valve repair, performed in our center. By doing this, the investigators want to evaluate predictors of outcome after repair.

ELIGIBILITY:
Inclusion Criteria:

* tricuspid valve insufficiency

Exclusion Criteria:

* younger than 18 years
* associated valvular surgery

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing isolated tricuspid valve repair
Sampling Method: Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2012-03-19 (Actual); Primary Completion 2012-06-30 (Actual); Study Completion 2013-03-01 (Actual)

PRIMARY OUTCOMES:
mortality | 10 year
Redo surgery | 10 year

SECONDARY OUTCOMES:
functional capacity assessed by CPET | 10 year
Atrial fibrillation | 10 year
Hospitalisation | 10 year
  hospitalisation for cardiovascular reasons
Functional capacity assessed by NYHA functional class | 10 years

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals Leuven, Leuven, Vlaams-Brabant, Belgium